CLINICAL TRIAL: NCT00278395
Title: A Phase II, Pharmacokinetic and Biologic Correlative Study of Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Advanced Renal Cell Carcinoma (RCC)
Brief Title: Vorinostat in Treating Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00087; NCI-2009-00087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000456500 (Other: Institute for Drug Development); #04-10 (Other: Institute for Drug Development); 6825 (Other: CTEP); U01CA069853 (NIH)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Vorinostat

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat (SAHA) twice daily on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Patients may have the option of continuing treatment beyond 52 weeks at the discretion of the investigator.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Given orally
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with advanced kidney cancer. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of vorinostat (SAHA), in terms of objective response and progression rate, in patients with advanced renal cell carcinoma.

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of this drug, in terms of toxicity profile, in these patients.

II. Evaluate overall survival, progression-free survival, and survival rate at 12 months in patients treated with this drug.

III. Correlate changes in biologic measurements with outcomes of patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral vorinostat (SAHA) twice daily on days 1-3, 8-10, 15-17, and 22-24. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Patients may have the option of continuing treatment beyond 52 weeks at the discretion of the investigator.

After completion of study treatment, patients are followed within 1 month and then approximately every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced renal cell carcinoma that is either metastatic or inoperable
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Disease is recurrent or refractory to interleukin-2 (IL-2) or interferon-based therapy OR new diagnosis in previously untreated patients who are not appropriate candidates to receive IL-2 based treatment
* Patients who have failed up to 4 lines of prior immunotherapy or biological therapy allowed
* No known brain metastases or leptomeningeal disease
* Stable brain metastases or curatively resected brain metastases without neurologic dysfunction for ≥ 6 months allowed
* ECOG performance status 0-2 OR Karnofsky 70-100%
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance > 50 mL/min
* Total bilirubin within normal limits
* AST/ALT ≤ 2.5 times ULN (≤ 5 times ULN if liver metastasis is present)
* No history of active malignancy (other than renal cell carcinoma) within the past 3 years other than nonmelanomatous skin cancer, in situ breast cancer, or in situ cervical cancer
* No history of allergic reactions to compounds of similar chemical or biological composition to vorinostat (SAHA)
* No uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No clinically significant hypercalcemia
* No significant traumatic injury within the past 21 days
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No gastrointestinal disease resulting in an inability to take oral medication
* No requirement for IV alimentation
* No active peptic ulcer disease
* Recovered from prior therapy
* Prior nephrectomy or resection of metastatic lesions allowed provided full surgical recovery has occurred
* No chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin)
* No radiotherapy within the past 4 weeks
* No valproic acid for at least 2 weeks prior to study enrollment
* No prior surgical procedures affecting absorption
* No major surgery within the past 21 days
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, Principal Investigator — Institute for Drug Development
Locations (2):
- United States (2):
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Institute for Drug Development, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open to recruitment on 12/5/2005, closed to recruitment on 3/3/09 at The University of Texas Health Science Center San Antonio at Cancer and Therapy Research Center
Groups:
- Vorinostat: The oral dose of vorinostat capsules was 300 mg two times a day for 3 consecutive days every week for 4 weeks, which constitutes on cycle of treatment. Treatment will be administered on an outpatient basis.
Period: Overall Study
Arm/Group | Vorinostat
Started | 14
Completed | 11
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Nonevaluable | 1

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat: The dose of vorinostat was 300 mg two times a day on the first 3 days of every week on a 4-week cycle.
Arm/Group | Vorinostat
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Objective response is measured using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST criteria.
  Complete Response (CR) - Disappearance of all target lesions, Partial Response (PR) - at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, Progressive Disease (PD) - At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, Stable Disease (SD) - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 1 year
Population: The overall duration of response will be estimated using the Kaplan-Meier method for all patients who presented with an objective response.
Measure: Number; unit: participants
Groups:
- Vorinostat: The dose of Vorinostat was 300 mg BID on the first 3 days of every week on a 4-week cycle. Dose reduction was allowed for adverse events (AE). Treatment was planned until disease progression (PD), death, unacceptable toxicity, or consent withdrawal.
Arm/Group | Vorinostat
Number analyzed (Participants) | 11
participants
  Best Objective Response Rate (ORR) | 4
  Progressive Disease | 7

2. Secondary Outcome: Progression-free Survival
Time Frame: 1 year
Population: Data were not collected
Groups:
- Progression Free Survival: No measurement reported
Arm/Group | Progression Free Survival
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS) and Median OS
Time Frame: 1 year
Population: Data were not collected
Groups:
- Overall Survival (OS) and Median OS: No measurement reported
Arm/Group | Overall Survival (OS) and Median OS
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Tolerability
Time Frame: 1 year
Population: Data were not collected
Groups:
- Safety and Tolerability: No participants measured
Arm/Group | Safety and Tolerability
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=14)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=14)
Nausea (Gastrointestinal disorders) | 7 (7)
Fatigue (Blood and lymphatic system disorders) | 7 (7)
Weight loss (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less